CLINICAL TRIAL: NCT05532774
Title: Efficacy and Safety of Defocusing Frame Glasses With Artificial Intelligence in Children and Adolescents Controlling Myopia Progression: A Multicenter, Randomized, Parallel-Controlled Clinical Trial
Brief Title: Efficacy and Safety of Defocusing Frame Glasses With Artificial Intelligence in Controlling Myopia Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kjb-ljkjj-v1.1-20220814
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ordinary defocusing frame glasses group (No Intervention): wear ordinary defocusing frame glasses
- AI defocusing frame glasses group (Experimental): wear defocusing frame glasses with artificial intelligence
  Interventions: Device: AI defocusing frame glasses

INTERVENTIONS:
Device: AI defocusing frame glasses — AI defocusing frame glasses have the function of eye behavior management, which can delay the progression of myopia through scientific management of eye behavior including outdoor light exposure (≥2 hours/day), duration of continuous close eye use (30 seconds rest every 30 minutes) and close eye distance (one punch, one foot and one inch), etc.
  Arms: AI defocusing frame glasses group

SUMMARY:
Background: Myopia refers to the pathological state in which the external parallel light enters the eye and focuses in front of the retina, resulting in the inability to clearly image on the retina. The number of myopia in China ranks first in the world. According to statistics from the National Health and Health Commission, the myopia rate of children and adolescents nationwide in 2020 will be as high as 52.7%. High myopia often leads to permanent visual impairment and even blindness. Retinopathy complicated by high myopia has become the first irreversible blinding eye disease in Shanghai and other regions. The problem is severe. Therefore, it is necessary to actively seek effective myopia treatment and correction methods to slow down the progression of myopia and the excessive extension of the eye axis and reduce the occurrence of complications.

Objective： On the basis of previous research, this study put forward the hypothesis that if behavior management (including outdoor light exposure and close-range eye-use behavior) can be strengthened in children with myopia wearing defocusing frame glasses, it is possible to achieve more effective myopia control effect, thereby not only ensuring safety also effectiveness. A randomized controlled clinical trial is conducted to evaluate the efficacy and safety of defocusing frame glasses with artificial intelligence in controlling myopia progression in children and adolescents.

Intervention: Group 1 ( AI defocusing frame glasses group), Group 2 ( Ordinary defocusing frame glasses group). The study period will be 2 years and each participant will be followed up every six month.

ELIGIBILITY:
Inclusion Criteria:

* The cycloplegic refraction of two eyes is [-0.50D, -5.0D) the astigmatism is ≥ -1.50D; or the cycloplegic refraction of either eye is [-5.00, -10.00D), the astigmatism is ≥ -2.50D;
* Willingness to wear only trial-provided defocusing frame glasses during the trial
* Have normal thinking and language communication skills, and be able to actively cooperate with the treatment as required;
* Written informed consent of guardian and child.

Exclusion Criteria:

* Allergy or intolerance to cycloplegic drugs;
* The anisometropia is greater than 1.50D;
* Using atropine, rigid orthokeratology lenses, bifocal lenses or progressive lenses, red light, acupuncture, etc. for myopia treatment;
* Strabismus/Amblyopia;
* History of eye surgery (including strabismus correction);
* Ocular or systemic diseases that may be related to the development of myopia or myopia: such as Marfan syndrome, neonatal retinopathy, diabetes, etc.;
* Corneal, conjunctival or eyelid damage or other diseases (keratoconus, herpes simplex keratitis, etc.);
* There are anatomical or skin factors that affect the wearing of spectacles;
* Other circumstances that the investigator judges inappropriate to participate in the trial.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-09-12 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
changes of spherical equivalent | at least 2 years
  Spherical equivalent as measured by cycloplegia autorefraction

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Eye Diseases Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang HY, Lam CSY, Tang WC, Leung M, To CH. Defocus Incorporated Multiple Segments Spectacle Lenses Changed the Relative Peripheral Refraction: A 2-Year Randomized Clinical Trial. Invest Ophthalmol Vis Sci. 2020 May 11;61(5):53. doi: 10.1167/iovs.61.5.53. PMID 32460315